CLINICAL TRIAL: NCT03807856
Title: Treating Acute Pancreatitis With Dabigatran, a Pilot Study
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Difficult recruitment
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Yan Bi, Principal Investigator, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-004345
Record Dates: First submitted 2019-01-15; First posted 2019-01-17 (Actual); Last update posted 2022-09-01 (Actual); Status verified 2022-08

CONDITIONS: Acute Pancreatitis
MeSH Terms: conditions — Pancreatitis | interventions — Dabigatran; Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dabigatran Etexilate Mesylate (Active Comparator): Dabigatran 150mg BID for 3 days
  Interventions: Drug: Dabigatran Etexilate Mesylate; Other: Standard of Care
- Standard of Care (Active Comparator): Standard treatment for acute pancreatitis
  Interventions: Other: Standard of Care

INTERVENTIONS:
Drug: Dabigatran Etexilate Mesylate — Dabigatran 150mg BID for 3 days
  Other Names: Pradaxa
  Arms: Dabigatran Etexilate Mesylate
Other: Standard of Care — Daily vital signs, lab work and one outpatient clinic visit

SUMMARY:
Researchers are studying the safety and efficacy of Dabigatran in the treatment of acute pancreatitis.

DETAILED DESCRIPTION:
Subjects with acute pancreatitis who meet the inclusion and exclusion criteria for the study will be recruited. Subjects will be randomized to receive either Dabigatran 150mg daily for three days or standard treatment. Vital signs, CBC, inflammatory markers and BMP, and bleeding complications will be evaluated daily for the next 7 days of until discharge whichever is sooner.

ELIGIBILITY:
Inclusion Criteria:

* Acute Pancreatitis (presence at least two of three features: typical pain, amylase or lipase >3 times UNL and AP on images)
* 18-75 years old
* Willingness to sign the informed consent
* Symptom onset within 72 hours

Exclusion Criteria:

* Under 18 years of age or over 75 years of age
* Pregnancy or lactating
* Presence of pseudo aneurysm on CT
* Predicted severe acute pancreatitis
* Unwilling or unable to sign the informed consent
* Had recent surgery or sphincterotomy
* Active pathological bleeding
* Concurrent use of anti-coagulation
* Known serious hypersensitivity reaction to Dabigatran
* CrCI <30mL/min or on dialysis
* Mechanical prosthetic valves
* Liver disease
* Cancer
* On Chemotherapy or immunosuppressant
* Persistent ALT, AST, Akl Phos >2 x ULN
* Active hepatitis C, active hepatitis B, and active hepatitis A
* Anemia (hemoglobin <10g/dL)
* Thrombocytopenia
* Concomitant use of P-gp inhibitors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2019-06-24 (Actual); Primary Completion 2020-07-23 (Actual); Study Completion 2020-07-23 (Actual)

PRIMARY OUTCOMES:
Adverse Events | One year
  Number of Reported Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yan Bi, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo clinic, Jacksonville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials